CLINICAL TRIAL: NCT00600262
Title: Efficacy of Intravitreal Bevacizumab for Severe Nonproliferative and Proliferative Diabetic Retinopathy.
Brief Title: Intravitreal Bevacizumab for Diabetic Retinopathy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-004
Record Dates: First submitted 2006-06-29; First posted 2008-01-24 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Severe Nonproliferative; Proliferative Diabetic Retinopathy; Active Photocoagulated Diabetic Retinopathy
Keywords: severe nonproliferative; proliferative diabetic retinopathy; active photocoagulated diabetic retinopathy; intravitreal bevacizumab

INTERVENTIONS:
Drug: intravitreal bevacizumab

SUMMARY:
Background: to evaluate the 3-month efficacy of a single dose of intravitreal bevacizumab on the progression of severe non proliferative diabetic retinopathy, proliferative diabetic retinopathy and active photocoagulated diabetic proliferative by evaluation of ischemic areas and regression of retinal and disc neovasculrization.

Methods: 40 patients were enrolled in a prospective, interventional study. Patients were treated with intravitreal bevacizumab 0.1ml (0.25mg). We evaluated visual acuity, neovascularization leakage points, capillary closure ischemic areas and macular edema by clinical examination and fluorescein angiography. A clinical examination was performed at baseline and days 1,14 and 30. Active leakage points were measured by fluorescein angiography at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Severe nonproliferative
* Proliferative diabetic retinopathy
* Active photocoagulated diabetic retinopathy

Exclusion Criteria:

* Previous vascular occlusion
* Glaucoma
* Uncontrolled hypertension, thromboembolic event
* Renal abnormalities
* Recent or planned surgery
* Coagulation abnormalities
* Panretinal photocoagulation of less than one month before
* Patients with known serious allergies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-12; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reyna-Castelan, MD, Principal Investigator — Asociación para evitar la ceguera en Mexico; Mariana Martinez-Castellanos, MD, Study Chair — Asociación para Evitar la Ceguera en México
Locations (1):
- Elizabeth Reyna Castelan, Mexico City, Mexico